CLINICAL TRIAL: NCT06729086
Title: Propofol vs Sevoflurane in Cardiac Surgery: a Randomized Clinical Trial During the Peroperative and Postoperative Phase
Brief Title: Propofol vs Sevoflurane in Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEHDF2230
Record Dates: First submitted 2024-09-27; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Complications; Cardiac Surgery; Neurologic Complications; Respiratory Complications
Keywords: propofol vs sevoflurane in cardiac surgery; peroperative; postoperative; randomized clinical trial; complications

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sedation using propofol (Placebo Comparator): this group will include all patients who will receive propofol during the cardiac surgery and afterwards in the intensive care unit during the post operative phase
  Interventions: Drug: sedation using propofol
- sedation using sevoflurane (Active Comparator): this group will include all patients who will receive sevoflurance druing the cardiac surgery and afterwards in the intensive care unit during the postoperative phase
  Interventions: Drug: sedation using sevoflurane

INTERVENTIONS:
Drug: sedation using propofol — The different complications studied will be for example respiratory, neurologic and cardiac based on several clinical and biological parameters.
  Arms: sedation using propofol
Drug: sedation using sevoflurane — The differents complications studied will be for example respiratory, neurologic and cardiac based on severl clinical and biological parameters.
  Arms: sedation using sevoflurane

SUMMARY:
The hypothesis of our study: presence of a relationship between the type of anesthesia and complications after cardiac surgery. The aim is to assess the benefit of using intravenous or inhaled anesthesia on the patients' stay and its complications.

DETAILED DESCRIPTION:
Cardiac surgery presents unique challenges for anesthesiologists as they are responsible for amnesia, analgesia, muscle relaxation, and maintenance of organ functions in the context of CPB-induced pathophysiological changes. Postoperative complications are vast and varied, leading to a prolonged stay in cardiac intensive care. However, the question of the superiority of one anesthesia protocol over another in cardiac surgery is debated.

The AHA (American Heart Association) recommended the use of inhalation anesthesia to reduce the risk of perioperative myocardial ischemia and infarction in 2011. However, in 2019, this recommendation lost a step in its level of proof and therefore the debate is still open.

Indeed, a "MYRIAD" study carried out on five continents determined that the administration of a halogenated volatile agent provided clinical benefit to patients undergoing coronary revascularization surgery. The study was randomized, single-blind, multicenter, carried out on patients scheduled for coronary bypass surgery with or without extracorporeal circulation (ECB).

Volatile halogenated agents (AVH) have cardioprotective properties via a pre- and post-conditioning phenomenon. Several meta-analyses have shown a benefit from the use of AVH during coronary surgery and in particular a reduction in mortality.

Note that the choice of type of anesthesia is made according to the habits of the department and the anesthetist and is in no way linked to the patient's condition or the intervention.

Given that within the HDF, there is an operating room and an intensive care unit dedicated to cardiac surgery forming an expertise and reference cell in Lebanon, it would be logical to introduce this sedation technique in order to establish new national recommendations and to report the Lebanese experience internationally. The ultimate goal is to provide the patient with optimal perioperative care.

The hypothesis of our study is that there is a relationship between the type of anesthesia and complications after cardiac surgery.

A prospective single-center randomized study targeting patients admitted to cardiovascular and thoracic intensive care for cardiac surgeries (PAC and valve replacement) at the Hôtel-Dieu de France, with the aim of evaluating the benefit of using intravenous anesthesia or inhaler on the patient stay and its complications. Two groups of patients will be formed respecting common characteristics in each group. Each sample of 50 patients will receive one type of anesthesia. All cases meeting the inclusion criteria mentioned below and spanning from 2023 to 2024 will be included in this study. Data collection will be done from the files of the patients concerned during their stay in the hospital intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* all patients above 18 yeras old that will undergo a cardiac surgery

Exclusion Criteria:

* below 18 yeras old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-04 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
determine the relationship between myocardial protection and type of anesthesia | 48 hours after the surgery
  troponin T dosage

SECONDARY OUTCOMES:
Association between the type of anesthesia and the speed of awakening | 48 hours after the surgery
  time taken to respond to simple commands, time elapsed to resume spontaneous ventilation
Association between the length of stay in intensive care and the type of anesthesia | 72 hours after the surgery
  duration of mechanical ventilation,
Determine a relationship between the type of anesthesia and the hemodynamic profile | 48 hours after the surgery
  measure cardiac output, vascular and pulmonary resistance, need for vasoamines
Association between the type of anesthesia and pulmonary complications | 72 hours after the surgery
  pulmonary complications: atelectasis, pneumonia, use of mechanical ventilation
Association between the type of anesthesia and neurological complications | 72 hours after the surgery
  early and late strokes, confusion, late and early strokes

IPD SHARING:
Plan to Share IPD: No